CLINICAL TRIAL: NCT00051402
Title: Phytoestrogens and Cognition in Menopause
Brief Title: Phytoestrogens and Memory Decline in Menopause
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000567-01A1 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-15 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Memory Loss; Postmenopause
Keywords: Postmenopausal; Memory Loss; Cognition; Phytoestrogens
MeSH Terms: conditions — Memory Disorders | interventions — Isoflavones

INTERVENTIONS:
Drug: Isoflavones

SUMMARY:
The purpose of this study is to investigate whether soy-derived phytoestrogens taken as dietary supplements improve memory function in postmenopausal women who have experienced early memory decline.

DETAILED DESCRIPTION:
Accumulating data has indicated that estrogens mediate enhancing effects on cognition and mood and may play a prophylactic role against age- and disease-related cognitive-cerebral decline. Phytoestrogens are plant-derived substances that have demonstrated estrogenic activity, but there is little prospective research regarding their effects on mental function. Mental health practitioners generally do not prescribe phytoestrogens. However, many women experiencing peri- and post-menopausal symptoms use marketed phytoestrogens under the perception of general health benefits, including presumably enhanced mental function. The purpose of this study is to develop preliminary data regarding the efficacy of isoflavone phytoestrogens in improving cognitive function in late middle-aged and elderly postmenopausal women with symptoms of memory impairment.

Participants in this study will be randomized to receive either isoflavone supplementation or placebo. The study will last for 16 weeks, during which participants will take the supplement pill or placebo three times a day. Participants will be assessed at study entry and at Week 16 for changes in basal cortisol levels, mood, and neuropsychological measures of executive function ability and episodic memory.

ELIGIBILITY:
Inclusion Criteria

* Postmenopausal women
* Mild memory or cognitive decline that does not meet the criteria for probable dementia

Exlcusion Criteria

* Hormone replacement therapy within 2 months prior to study entry
* Psychiatric medications within 30 days prior to study entry

Min Age: 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2002-12; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krikorian, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States